CLINICAL TRIAL: NCT06839716
Title: Prospective Randomized Controlled Study of Ropivacaine-Poloxamer 407 Based Gel Application and TAP Block for Postoperative Pain Management Following Laparoscopic/Robotic Gastrectomy
Brief Title: Comparison of Ropivacaine-Poloxamer 407 Hydrogel and TAP Block for Postoperative Pain Management in Laparoscopic/Robotic Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2024-0451
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine-Poloxamer 407 hydrogel group (Experimental): Patients withRopivacaine-Poloxamer 407 hydrogel applied to the peritoneal and subcutaneous layers at the incision site.
  Interventions: Procedure: Arm I (Ropivacaine-Poloxamer 407 hydrogel group)
- TAP block group (Active Comparator): Patients with Ultrasound-guided subcostal TAP block with 0.375% ropivacaine (15 mL per side).
  Interventions: Procedure: Arm II (TAP block group)

INTERVENTIONS:
Procedure: Arm I (Ropivacaine-Poloxamer 407 hydrogel group) — Patients receive intraoperative application of Ropivacaine-Poloxamer 407 hydrogel at the incision site. A mixture of 0.75% Ropivacaine (22.5 mg, 3 mL) and Poloxamer 407-based gel (Welpass, 6 mL) is prepared. The hydrogel is applied as 4 mL between the peritoneum and fascia, and 2 mL is injected subcutaneously around the incision before skin closure. This intervention aims to provide sustained local anesthesia for up to 72 hours.
  Arms: Ropivacaine-Poloxamer 407 hydrogel group
Procedure: Arm II (TAP block group) — Patients undergo ultrasound-guided subcostal transversus abdominis plane (TAP) block before anesthesia emergence. A total of 30 mL of 0.375% Ropivacaine (15 mL per side) is injected bilaterally between the internal oblique and transversus abdominis muscles. TAP block is a regional anesthesia technique known for effective postoperative pain control, typically lasting 24 to 48 hours.
  Both groups receive standardized postoperative analgesia, including IV acetaminophen, fentanyl via patient-controlled analgesia (PCA), and rescue pethidine as needed.
  Arms: TAP block group

SUMMARY:
This study aims to determine whether Ropivacaine-Poloxamer 407 hydrogel provides non-inferior pain control compared to TAP block for patients undergoing minimally invasive gastrectomy. The results will guide postoperative pain management practices and enhance recovery protocols for gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically confirmed diagnosis of gastric adenocarcinoma prior to surgery.
2. Patients who have undergone a complete surgical resection (R0 resection).
3. Patients with an ASA (American Society of Anesthesiologists) score of 3 or below.
4. Patients aged 20 years or older.
5. Patients who have undergone laparoscopic or robotic gastrectomy

Exclusion Criteria:

1. Patients under 19 years of age.
2. Presence of ascites or peritoneal metastasis.
3. Patients who have undergone preoperative chemotherapy or radiotherapy.
4. Diagnosis of malignancies other than gastric cancer.
5. Uncontrolled diabetes, autoimmune diseases, hypertrophic scars, or keloid history affecting wound healing.
6. History of allergy or adverse reactions to Ropivacaine or other local anesthetics.
7. Pregnant women.
8. Patients with preoperative chronic pain conditions, including CRPS.
9. Patients with long-term preoperative use of opioid analgesics.
10. Patients with psychiatric disorders deemed likely to interfere with study participation.
11. Patients with severe liver disease, renal disease, or arrhythmia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total fentanyl consumption within 72 hours postoperatively. | Over the first 72 hours after surgery.
  The total amount of fentanyl administered to the patient via IV PCA during the initial 72-hour postoperative period will be recorded and compared among groups to assess analgesic efficacy.

SECONDARY OUTCOMES:
Fentanyl usage at 12, 24, 48 hours. | Fentanyl usage at 12, 24, 48 hours.
  Pain intensity: Numerical Rating Scale (NRS) scores ranging from 0 (no pain) to 10 (worst pain) assessed both at rest and during movement.
NRS pain scores at 24, 48, and 72 hours (at rest and during movement). | NRS pain scores(0-10 / 0: no pain / 10: worst pain) at 24, 48, and 72 hours (at rest and during movement).
  Bowel function: Time to resume normal gastrointestinal activity.
Pethidine usage at 24, 48, 72 hours | Pethidine usage at 24, 48, 72 hours
  PONV: Incidence of nausea and vomiting documented along with severity scores.
Time to first flatus and bowel movement. (up to 1 month) | 1 month
  The time from surgery completion to the first passage of gas and bowel movement will be recorded to assess postoperative gastrointestinal recovery.
Incidence of seroma or surgical site infection. (up to 1 month) | 1 month
  The presence of seroma or surgical site infection (SSI) will be evaluated through clinical examination and recorded according to standardized criteria.
Quality of Recovery (QoR-15) scores at baseline and 72 hours | 72 hours postoperatively
  Quality of recovery will be assessed using the 15-item Quality of Recovery (QoR-15) questionnaire, which evaluates physical comfort, emotional state, and overall well-being.(Quality of Recovery (QoR-15) score 0-10 on each items/ 0: worst recovery / 10: best recovery)
Peak Cough Flow (baseline and 72 hours) | Baseline (preoperatively) and 72 hours postoperatively
  Peak cough flow (PCF) will be measured using a peak flow meter to assess respiratory function and recovery after surgery.
Length of hospital stay. (up to 1 month) | up to 1 month
  The total number of days from surgery to hospital discharge will be recorded to evaluate recovery speed and efficiency.
Incidence of postoperative nausea and vomiting (PONV). (up to 72 hours) | 72 hours postoperatively
  The occurrence of postoperative nausea and vomiting (PONV) will be documented, and severity will be assessed using a standardized scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided